CLINICAL TRIAL: NCT03089411
Title: Collection of Additional Data Followed the Study "A Phase III Study of Velcade (Bortezomib) Thalidomide Dexaméthasone (VTD) Versus Velcade (Bortezomib) Cyclophosphamide Dexaméthasone (VCD) as an Induction Treatment Prior to Autologous Stem Cell Transplantation in Patients With Newly Diagnosed Multiple Myeloma"
Brief Title: Collection of Additional Data Followed the Study IFM 2013-04
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC13_0284_03
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Myeloma Multiple
Keywords: myeloma multiple; newly diagnosed
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Collection of retrospective additional data (survival, biological, disease response data) following the study IFM 2013-04.

ELIGIBILITY:
Patients newly diagnosed with symptomatic Multiple Myeloma (MM) patient

1. - 18 ≤ age < 66 years
2. - Eastern Cooperative Oncology Group Performance Status of 0, 1 or 2
3. - Patients must be eligible for Autologous Stem Cell Transplantation
4. - Patients must have measurable disease by serum M-protein ≥ 10 g/L and/or urine M-protein ≥200mg/day
5. - Female patients of child-bearing potential (FCBP):

   * Must agree to have medically supervised pregnancy tests prior to starting study and every 21 days, including 4 weeks after the end of study treatment. This applies even if the patient practices complete and continued sexual abstinence.
   * Must agree to use and be able to comply with effective contraception without interruption, 28 days prior to starting study drug, during the study therapy (including during periods of dose interruptions), and for 28 days after discontinuation of study therapy.
6. - Male Patients:

   * Must agree to use a condom during sexual contact with a FCBP, throughout study drug therapy, during any dose interruption and for one week after discontinuation of study therapy
   * Must agree to not donate semen during study drug therapy and for one week after discontinuation of study therapy
7. - All patients must:

   * Agree to abstain from donating blood while taking study drug therapy and for one week after discontinuation of study drug therapy
   * Agree not to share study medication with another person.
8. - Patients must be capable of giving informed consent
9. - Patients must be affiliated with French social security system

Exclusion Criteria:

1. - Asymptomatic Multiple myeloma
2. - Non-secretory Multiple myeloma
3. - Proven AL-amyloidosis
4. - Age ≥ 66 years old
5. - Prior or current systemic therapy for Multiple myeloma, including steroids (except for emergency use of a 4-day block of dexamethasone before randomization, maximum total dose allowed 160 mg)
6. - Radiation therapy in the 2 weeks preceding randomization
7. - National Cancer Institute grade ≥ 2 peripheral neuropathy
8. - Haemoglobin < 8g/dL
9. - Absolute neutrophil count < 1,000 cells / µL, platelet count < 50,000 cells / µL
10. - Creatinine level > 170 µmol/L or requiring dialysis.
11. - Bilirubin, transaminases or GamaGT > 3 UNL (upper normal limit)
12. - Positive HIV serology, evidence of active Hepatitis B and C infection
13. - Severe active infection
14. - Inability to comply with an anti-thrombotic treatment regimen
15. - A personal medical history of severe psychiatric disease
16. - Uncontrolled diabetes contraindicating the use of high-dose dexamethasone
17. - Non-controlled or severe cardiovascular disease (including a myocardial infarction in the 6 months prior to recruitment)
18. - A personal medical history of cancer unless the patient has been without relapse after treatment discontinuation > or = 5 years (except for basocellular skin cancer or in situ cervical cancer)
19. - Use of any investigational drug in the 30 days preceding randomization 22 - Pregnant or lactating women. 23 - Adults under juridical protection 24 - Known or suspected hypersensitivity to any of the study therapies or excipients 25 - Necessity of vaccination for yellow fever or with any other live vaccines

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 340 patients newly diagnosed with symptomatic Multiple Myeloma (MM) patient included in the study IFM 2013-04
Sampling Method: Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-07-15 (Estimated); Study Completion 2017-07-15 (Estimated)

PRIMARY OUTCOMES:
Number of death | 6 months
  To evaluate Overall and Progression-Free Survival

CONTACTS AND LOCATIONS:
Locations (62):
- France (62):
  - Centre Hospitalier de la région d'Annecy, Annecy, Pringy,
  - CHRU Hôpital Sud, Amiens
  - CHU Angers, Angers
  - Centre Hospitalier Argenteuil, Argenteuil
  - Centre Hospitalier H.Duffaut, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHRU de Besançon, Besançon
  - Hôpital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre hospitalier Pierre Oudot, Bourgoin
  - Hôpital A.Morvan, Brest
  - CHU Caen Côte de Nacre, Caen
  - CH René Dubos, Cergy-Pontoise
  - Centre Hospitalier William Morey, Chalon/saone
  - Hôpital d'instruction des armées Percy, Clamart
  - CHU d'Estaing, Clermont-Ferrand
  - Hôpitaux civils de Colmar, Colmar
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - CHRU Dijon, Dijon
  - Centre Hospitalier Général, Dunkirk
  - CHRU - Hôpital A.Michallon, Grenoble
  - Centre hospitalier départemental Vendée, La Roche-sur-Yon
  - Hôpital Louis Pasteur, Le Coudray
  - Centre Jean Bernard, Le Mans
  - CH Le Mans, Le Mans
  - Hopital Saint Vincent de Paul, Lille
  - CHRU - Hôpital Claude Huriez, Lille
  - CHU de Limoges, Limoges
  - Hôpital Du Scorff, Lorient
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - CHR Metz Thionville, Metz
  - Centre Hospitalier intercommunale Meulan les mureaux, Meulan-en-Yvelines
  - Hopital E Muller, Mulhouse
  - Nantes University Hospital, Nantes
  - Hôpital de l'Archet 1, Nice
  - Groupe Hospitalo-Universitaire Carémeau, Nîmes
  - Institut CURIE, Paris
  - Hôpital Cochin, Paris
  - CHU - Hôpital St-Antoine, Paris
  - Hôpital Pitié-Salpétrière, Paris
  - AP-HP Hôpital Necker, Paris
  - CH Saint Jean, Perpignan
  - CHRU - Hôpital du Haut Lévêque, Pessac
  - Centre Hospitalier de PERIGUEUX, Périgueux
  - Centre Hospitalier Lyon sud, Pierre-Bénite
  - CHRU - Hôpital Jean Bernard, Poitiers
  - Hôpital R.Debré, Reims
  - CHRU - Hôpital de Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Yves le Foll, Saint-Brieuc
  - Centre René Huguenin, Saint-Cloud
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Centre Hospitalier, Saint-Quentin
  - Centre hospitalier st Malo, St-Malo
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHRU - Hôpital Purpan, Toulouse
  - CHRU - Hôpital Bretonneau, Tours
  - CHRU - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique Vannes et Auray, Vannes